CLINICAL TRIAL: NCT01319500
Title: Drug Utilization Study on the Prescribing Indications for Yasmin® and Other OCs in Croatia
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG 2009_02
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-10

CONDITIONS: Contraception
Keywords: Drug Utilization; Oral Contraceptives

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Yasmin: Users of the drospirenone/ethinylestradiol (DRSP/EE) containing OC "Yasmin"
- Other OCs: Users of OCs except Yasmin ("Other OCs")

SUMMARY:
This study investigates the drug utilization pattern of Oral Contraceptives (OC) in Croatia. Gynecologists and Dermatologists were asked to contribute OC prescribing data to this study.

DETAILED DESCRIPTION:
Large, prospective non-interventional cohort studies with active surveillance of study participants indicate that many users of oral contraceptives use these preparations not only for contraception but also for the treatment of hormone-dependent diseases and symptoms - such as premenstrual dysphoric disorder, acne, endometriosis, ovarian cysts, polycystic ovary syndrome, bleeding disorders and painful periods. In the International Active Surveillance Study of Women Taking Oral Contraceptives (INAS) more than 30% of participants reported that they use their OC for contra¬ception as well as for the treatment of one of the mentioned conditions.

It is also conceivable that some women use OC not for contraception but only for one of these hormone-dependent conditions. In most instances the exclusive use for these conditions would constitute off-label use as only few preparations have a stand-alone approved indication for one of these conditions.

For many countries the actual extent of off-label use of OCs for these conditions is unknown. This applies also to Croatia. Therefore, the Croatian health authority requested a drug utilization study to investigate current prescribing indications for Yasmin® and other OCs in Croatia. The study details were agreed upon with the Croatian health authority.

ELIGIBILITY:
Inclusion Criteria:

* women with an OC prescription during the timeframe (Feb-March 2011)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Overall, a representative sample of 100 gynecologists and 31 dermatologists are asked to contribute OC prescribing data to this study.
Sampling Method: Probability Sample
Enrollment: 3776 (Actual)
Dates: Start 2009-02

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Dinger, MD, PhD, Principal Investigator — Berlin Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemiology and Health Research Berlin, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A representative sample of 100 Croatian gynecologists and 31 dermatologists were asked to fill in a questionnaire for each of their oral contraceptive (OC) prescriptions from February 16, 2009 to March 15, 2009. Questions included the name of the OC, date and reason for prescription, and the reproductive status and demographics of the patients.
Groups:
- Other OCs: Users of oral contraceptives (OCs) except Yasmin ("Other OCs")
Period: Overall Study
Arm/Group | Yasmin | Other OCs
Started | 1187 | 2589
Completed | 1187 | 2589
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Yasmin: Users of the DRSP/EE containing OC "Yasmin"
- Total: Total of all reporting groups
Arm/Group | Yasmin | Other OCs | Total
Number analyzed (Participants) | 1187 | 2589 | 3776
Age Continuous [Mean (Standard Deviation); unit: years] | 23.8 (5.0) | 26.5 (6.3) | 25.7 (6.0)
Age, Customized [Number; unit: participants]
  <18 years | 67 | 62 | 129
  >=18 and <40 years | 1097 | 2398 | 3495
  >=40 years | 11 | 79 | 90
  Missing | 12 | 50 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1187 | 2589 | 3776
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Croatia | 1187 | 2589 | 3776

OUTCOME MEASURES:

1. Primary Outcome: OC Prescriptions by Treatment Group and Prescribing Medical Specialists
Description: Prescriptions of Yasmin and Other OCs by different physicians (private gynecologists, public gynecologists and dermatologists)
Time Frame: February 2009 - March 2009
Measure: Number; unit: Prescribing physicians
Arm/Group | Yasmin | Other OCs
Number analyzed (Participants) | 1187 | 2589
Prescribing physicians
  Gynecologists (private practice) | 244 | 331
  Gynecologists (public practice) | 929 | 2213
  Dermatologists | 14 | 45

2. Primary Outcome: Reasons for OC Prescriptions
Description: The main reasons for OC prescription: contraception only; contraception combined with non-contraceptive reasons; non-contraceptive reasons only.
Time Frame: February 2009 - March 2009
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Yasmin | Other OCs
Number analyzed (Participants) | 1187 | 2589
percentage of participants
  Contraception only | 53.8 [51.0 to 56.7] | 57.8 [55.9 to 59.7]
  Contraception plus non-contraceptive reasons | 38.8 [36.0 to 41.6] | 29.7 [27.9 to 31.5]
  Non-contraceptive reasons only | 5.2 [4.0 to 6.7] | 11.6 [10.4 to 12.9]

3. Primary Outcome: Non-contraceptive Reasons for OC Prescriptions (Reported by Women Who Used OCs for "Contraceptive and Non-contraceptive" and "Non-contraceptive Only" Reasons
Description: Non-contraceptive reasons for OC prescriptions (including both categories: "contraception plus non-contraceptive reasons" and "non-contraceptive reasons only"
Time Frame: February 2009 - March 2009
Measure: Number; unit: number of participants
Arm/Group | Yasmin | Other OCs
Number analyzed (Participants) | 522 | 1068
number of participants
  Acne | 226 | 338
  Painful period | 212 | 246
  PCOS | 199 | 405
  Abnormal menstrual bleeding | 100 | 254
  Bleeding on demand | 63 | 177
  PMS | 59 | 130
  Ovarian cysts | 34 | 80
  Uterine disease | 33 | 47
  PMDD | 4 | 19
  Hyperandrogenism | 3 | 10
  Other | 0 | 3

4. Primary Outcome: Non-contraceptive Reasons for OC Prescriptions (Reported by Women Who Used OCs for Non-contraceptive Reasons Only)
Description: Exclusively non-contraceptive reasons for OC prescriptions (no contraception intended; category "non-contraceptive reasons only"
Time Frame: February 2009 - March 2009
Measure: Number; unit: number of participants
Arm/Group | Yasmin | Other OCs
Number analyzed (Participants) | 62 | 300
number of participants
  PCOS | 29 | 131
  Acne | 22 | 97
  Painful period | 15 | 40
  Abnormal menstrual bleeding | 8 | 94
  Bleeding on demand | 7 | 22
  PMS | 3 | 10
  Ovarian cysts | 5 | 17
  Uterine disease | 4 | 22
  PMDD | 0 | 1
  Hyperandrogenism | 0 | 4

5. Primary Outcome: Reasons for OC Prescriptions by Gynecologists and Dermatologists
Time Frame: February 2009 - March 2009
Measure: Number; unit: number of participants
Groups:
- Gynecologists (All): All gynecologists (private and public)
- Gynecologists (Private Practice Only): Gynecologists in private practice only
- Gynecologists (Public Practice Only): Gynecologists in public practice only
- Dermatologists: All dermatologists
- Total: All gynecologists (private and public) and dermatologists
Arm/Group | Gynecologists (All) | Gynecologists (Private Practice Only) | Gynecologists (Public Practice Only) | Dermatologists | Total
Number analyzed (Participants) | 3717 | 575 | 3142 | 59 | 3776
number of participants
  Contraception only | 2130 | 347 | 1783 | 5 | 2135
  Contraceptive plus non-contraceptive reasons | 1201 | 178 | 1023 | 27 | 1228
  Non-contraceptive reasons only | 337 | 32 | 305 | 25 | 362

ADVERSE EVENTS:
Description: Adverse event data were not collected.
Arm/Group | Yasmin | Other OCs
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No